CLINICAL TRIAL: NCT00458159
Title: A Phase I, Open-Label, Dose-Escalation Study of CC-11006 In Subjects With Low- or Intermediate-1 Risk Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The compound has a benign safety profile with short-term use, clinically sig efficacy responses have not been demonstrated, or if so, have not been sustained.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-11006-MDS-001
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Myelodysplastic Syndrome
Keywords: CC-11006; RA; MDS; Celgene; RCMD-RS; RARS; RAEB-1; Low-or Intermediate-1-Risk Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: CC-11006

INTERVENTIONS:
Drug: CC-11006 — Doses: 10mg, 15mg, 25mg, 35mg, & 50mg, taken once daily, orally.

SUMMARY:
A Phase I, Open-Label, Dose-Escalation Study of CC-11006 In Subjects With Low- or Intermediate-1 Risk Myelodysplastic Syndromes.

ELIGIBILITY:
Study Population Key Inclusion Criteria

* Age greater than 18 years.
* Able to understand and voluntarily sign an informed consent form.
* A diagnosis of de novo myelodysplastic syndrome (MDS) of at least 12 weeks duration, with one of the following subtypes (See WHO Classification and Criteria for Myelodysplastic Syndromes).

  1. Refractory anemia (RA)
  2. Refractory cytopenia with multilineage dysplasia (RCMD)
  3. Refractory anemia with ring sideroblasts (RARS)
  4. Refractory cytopenia with multilineage dysplasia and ringed sideroblasts (RCMD-RS)
  5. Refractory anemia with excess blasts (RAEB-1 [5-9% blasts])
  6. RAEB-2 (10%-19% blasts)
  7. MDS-Unclassified (MDS-U)
  8. MDS with chromosome 5q deletion (MDS 5q-)
* At least two hemoglobins < 9 g/dL (untransfused) or transfusion-dependence defined as requiring at least 4 units of RBCs in the 56 days prior to Study Day 1 (start of CC-11006 treatment).
* Tried and failed one or more conventional first-line treatments for MDS with anemia including Revlimid®, recombinant erythropoietins, 5-azacitidine, decitibine or other associated therapies.
* More than 28 days (from Study Day 1) must have elapsed since any previous treatment (including Revlimid®) for MDS with anemia, other than transfusion(s).
* An ECOG Performance status of 0, 1 or 2 • Able to adhere to the study visit schedule and other protocol requirements.
* Females of childbearing potential (FCBP)† must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse for at least 28 days before starting study drug, while on study drug, during dose interruptions, and 28 days after the last dose of study drug. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device, hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods, if needed.

Before starting study drug:

* FCBP must have two negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to starting study drug. The first test must be performed within 10 - 14 days and the second negative pregnancy test within 24 hours prior to the start of study drug. The subject may not receive study drug until the Investigator has verified a negative pregnancy test.
* Will be counseled about pregnancy precautions, potential risks of fetal exposure.

Male Subjects:

* Must agree to use a latex condom during any sexual contact with females of childbearing potential during study drug treatment, during dose interruptions, and for at least 28 days following discontinuation of study drug even if they have undergone a successful vasectomy.
* Agree to abstain from donating semen or sperm while taking study drug and for 28 days after stopping study drug.

While on study and during dose interruptions:

* FCBP with regular cycles must agree to have pregnancy tests weekly for the first 28 days and then every 28 days while on study drug, during dose interruptions and at day 28 day following discontinuation of study drug. If menstrual cycles are irregular, the pregnancy testing must occur every 14 days.
* The subject may not receive study drug until the Investigator has verified a negative pregnancy test.
* No more than a 28-day supply of study drug is to be dispensed at a time.
* In addition to the required pregnancy testing, the Investigator must confirm with FCBP that they are continuing to use the two reliable methods of birth control at each visit.
* Counseling about pregnancy precautions must be done at a minimum of every 28 days. Subjects must be reminded of the potential risks of fetal exposure at each visit and to not share drug.
* Pregnancy testing and counseling must be performed if a subject missed her period or if there is any abnormality in her pregnancy test or in her menstrual bleeding. Study drug treatment must bediscontinued during this evaluation.
* Females must agree to abstain from breastfeeding while on study, during dose interruptions and for 28 days after last dose of study drug.

Male Subjects:

-Counseling not to share drugs, donate blood, sperm or semen, and on contraceptive use, including counseling on emergency contraception must be done at a minimum of every 28 days.

Upon discontinuation of study drug:

* Pregnancy test will be performed for FCBP at study termination and at day 28 after last dose of study drug.
* Females must agree to abstain from breastfeeding for 28 days after last dose of study drug.
* Male and FCBP subjects must follow all birth control requirements as those required while on study drug for 28 days after last dose of study drug.
* Both males and females must agree to abstain from donating blood or ova (for females) while taking study drug and for 28 days after stopping study drug.
* Males must not donate sperm or semen for 28 days after last dose of study drug.

If pregnancy does occur during treatment, study drug must be immediately discontinued. Key Exclusion Criteria

* Myelosclerosis (or myelofibrosis) occupying more than 30% of marrow space.
* Bone marrow blast ≥ 20 %.
* The following laboratory abnormalities:

  1. Absolute neutrophil count (ANC) < 500 cells/L (0.5 x 109/L)
  2. Platelet count < 50,000/L (50 x 109/L)
  3. Serum creatinine > 2.0 mg/dL (177 mol/L)
  4. Serum SGOT/AST or SGPT/ALT > 3.0 x upper limit of normal (ULN)
  5. Serum total bilirubin > 2 x the ULN secondary to hemolysis in the absence of any known intrinsic liver disease
* A history of active tuberculosis requiring treatment within the previous 3 years (of Study Day 1) or opportunistic infections, including but not limited to evidence of active cytomegalovirus, active Pneumocystis carinii, or atypical mycobacterium infection, etc., or documented HIV infection, within the previous 6 months (of Study Day 1). Subjects with evidence of an old tuberculosis infection without documented adequate therapy are also excluded.
* A history of active non-hematopoietic malignancy, or a similar diagnosis within 3 years of Study Day 1 (except basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ).
* A history of venous thromboembolism.
* Clinically significant anemia due to factors such as iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis or gastrointestinal bleeding (if a marrow aspirate is not evaluable for storage iron, transferrin saturation must be > 20 % and serum ferritin not less than 50 ng/mL).
* Any clinically significant pulmonary, cardiac, vascular, endocrine, hepatic, neurological, gastrointestinal or genitourinary disease unrelated to underlying hematological disorder.
* Any life-threatening or active infection requiring parenteral antibiotic therapy.
* Chromosome abnormalities common to de novo acute myelogenous leukemia (AML), i.e., t(8:21), t(15;17), and inv (16).
* Known hepatitis-B surface antigenemia or positive hepatitis-C antibodies.
* Known HIV-1 positivity.
* Greater than Grade 2 neuropathy.
* Any medical condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Any other serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Subjects who require ongoing treatment with corticosteroids.
* Use of cytotoxic chemotherapeutic agents or experimental agents (agents that are not commercially available) for the treatment of MDS within 28 days of the first day of study drug treatment.
* Recombinant human erythropoietin (rHuEPO) therapy within 28 days of the first day of study drug treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2008-10-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of CC-11006 | 2 cohorts

SECONDARY OUTCOMES:
Safety of CC-11006-MDS-001 | Ongoing basis

CONTACTS AND LOCATIONS:
Overall Officials: Alan List, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (7):
- United States (7):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York
  - Wake Forest University School of Medicine Bowman Gray Campus, Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Brandenburg N, et al. Venous thromboembolism in patients with myelodysplastic syndrome treated with lenalidomide: Incidence and risk factors. Presented at 2008 ASCO Annual Meeting, May 30-June 3, 2008, Chicago, IL. Abstract No. 7084.